CLINICAL TRIAL: NCT01436266
Title: Effect of Preoperative Buccal Misoprostol on Blood Loss in Second-trimester
Brief Title: Effect of Preoperative Buccal Misoprostol on Blood Loss in Second-trimester Dilation and Evacuation Abortion
Acronym: PreopMiso
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-30452
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Abortion; Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Misoprostol; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Misoprostol (Active Comparator): 400 mcg buccally 2 hours prior to procedure
  Interventions: Drug: Misoprostol
- Placebo (Folic acid) (Placebo Comparator): Two 1-mg tablets buccally 2 hours prior to procedure
  Interventions: Other: Folic acid

INTERVENTIONS:
Drug: Misoprostol — 400 mcg buccally 2 hours prior to procedure
  Other Names: Cytotec
  Arms: Misoprostol
Other: Folic acid — 2mg buccally 2 hours prior to procedure
  Other Names: Vitamin B9
  Arms: Placebo (Folic acid)

SUMMARY:
Misoprostol is a medication used extensively in obstetrics and gynecology for its ability to aid in softening the cervix as well as decreasing blood loss after abortion or vaginal delivery. Opinions vary as to its usefulness in aiding in cervical dilation, and in decreasing blood loss. The investigators propose to conduct a randomized, placebo-controlled trial to evaluate whether misoprostol given buccally 2 hours prior to second trimester surgical abortion decreases blood loss from the procedure. The investigators will also assess whether misoprostol improves cervical dilation, changes the length of the procedure, changes the need for additional mechanical dilation, changes the subjective ease of the procedure, and changes a woman's pain.

DETAILED DESCRIPTION:
This project is a placebo-controlled, double-blinded randomized controlled trial comparing the effect of misoprostol 400mcg buccally to placebo on blood loss in second trimester surgical abortion between 16-21 weeks gestation. The probability of group assignment is 50% with half of the women randomized to misoprostol and half to placebo (folic acid 1 mg).

Folic acid was chosen at the placebo as it looks similar to misoprostol, and when it is held in the cheek it has very little taste, similar to misoprostol. A compounded placebo that was tasteless had a very different appearance and was not suitable as a control.

Consent will be obtained after consent for the abortion has been completed and counseling and explanation of the abortion has been completed. Consent may be obtained before the abortion procedures have begun of the day prior to abortion (osmotic dilator placement and induction of fetal demise if appropriate), or after these procedures have been completed. No study procedures take place on the day prior to abortion.

On the day of the abortion, 1 hour prior to the procedure, the following study procedures will be conducted. Women will be given the study medication, which consists of two tablets of either misoprostol 200 mcg (400 mcg total) or placebo (folic acid 2 mg). The medication will be dispensed from opaque sequentially numbered vials so that double-blinding is maintained. The subject will be asked questions about symptoms prior to administration of the study medication. She will then hold the medication buccally (in her cheek) for 20 minutes and then swallow any remaining tablet. Immediately prior to the abortion, the subject will be asked about her symptoms again.

The abortion will commence 1 hour after administration of the study medication. The following study procedure will be done at the start of the abortion. The amount of cervical dilation will be measured by cervical dilators, starting with the largest dilator and progressively using smaller dilators until the largest one that will pass is determined. This generally takes less than 30 seconds.

The abortion will then be done with a combination of suction and extraction, which is part of standard clinical care at BMC. The following research procedures will be conducted: the length of the procedure will be recorded, and the woman will be asked afterward about her pain level during the abortion. This concludes the study procedures for the woman. Her time in the study is one day.

After the abortion, the fetus and placenta will be removed from the collected specimen and weighed and sent to pathology as per usual clinical procedure. The following study procedure will be done. The collected fluid from the suction machine, consisting of blood and amniotic fluid, will be measured. If the drapes or towels have been soiled with blood or fluid, they will be weighed and the amount added to the total measured from the suction machine. The amount of blood will be calculated by comparison with the expected amount of amniotic fluid as published by Hern (attached in Section S). Note that the amount of fetal blood is very small, less than 20 ml at the highest gestational age in this study, and will not appreciably change the total. If all of the blood and fluid has been collected into the suction jar (and none of the towels are soiled), then 5 ml of the mixed fluid will be sent for a hemoglobin level, and the percentage of blood calculated from that, as pure amniotic fluid will have a hemoglobin level of zero. This results will be used for confirmation when available, but will not be used as the primary outcome. Measurements on the fluid will be completed on the day of abortion. The fluid is normally discarded and will be discarded after measures are complete.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Gestational age between 16 weeks 6 days and 20 weeks 6 days gestation by ultrasound dating on the day of enrollment
* Ultrasound used for dating purposes must be within the last two weeks.
* Women 18-50 years of age undergoing surgical termination of pregnancy

Exclusion Criteria:

* Spontaneous fetal demise
* Ruptured membranes or intrauterine infection
* Fibroids that significantly distort the uterine shape
* Uterine abnormality such as unicornuate uterus
* Prior transmural myomectomy
* Severe oligohydramnios
* Morbid obesity with BMI>45
* Inability to place osmotic dilators

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Sonalkar, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible women will be identified by the clinician caring for the patient who will mention the study. If interested research staff will describe the study in detail and obtain consent from interested patients. The clinician who cares for the patient, and the physician who does the abortion procedure, will not be involved in the research procedures.
Pre-assignment Details: Three subjects were consented, one of which was ineligible after consent because she had spontaneous rupture of amniotic membranes prior to the abortion procedure. The other two subjects were enrolled.
Groups:
- Active Comparator: Misoprostol: 400 mcg buccally 2 hours prior to procedure
- Placebo Comparator: Placebo (Folic Acid): Two 1-mg tablets buccally 2 hours prior to procedure
Period: Overall Study
Arm/Group | Active Comparator: Misoprostol | Placebo Comparator: Placebo (Folic Acid)
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Misoprostol | Placebo Comparator: Placebo (Folic Acid) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Placebo Comparator: Placebo (Folic acid): Female | 1 | 1 | 2
  Placebo Comparator: Placebo (Folic acid): Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: 500 cc or more
Time Frame: one day following the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Misoprostol | Placebo Comparator: Placebo (Folic Acid)
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Misoprostol | Placebo (Folic Acid)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
1 of the 3 consented subjects became ineligible due to spontaneous rupture of amniotic membranes prior to the abortion. Early study termination, the PI left the institution, and study records could not be located for secondary data outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes